CLINICAL TRIAL: NCT01243450
Title: Bioequivalence Study of Generic Tretinoin 0.04% Microsphere Gel, 0.04% Retin-A Micro® and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spear Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAM-04
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2014-11

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active generic (Active Comparator): Treatment of acne for 12 weeks with generic tretinoin
  Interventions: Drug: Tretinoin
- Placebo (Placebo Comparator): Treatment of acne for 12 weeks with Placebo
  Interventions: Drug: placebo
- Brand (Active Comparator): Treatment of acne over 12 weeks with tretinoin Brand
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Tretinoin — Treatment of acne
  Other Names: active medication
  Arms: Active generic; Brand
Drug: placebo — treatment of acne
  Other Names: inactive medication
  Arms: Placebo

SUMMARY:
The objective will be to assess clinical bioequivalence of 0.1% Retin-A Micro® Gel and Spear Pharmaceutical's generic 0.1% Tretinoin Microsphere Gel with a placebo arm.

DETAILED DESCRIPTION:
Acne study

ELIGIBILITY:
A subject will be eligible to participate if they meet all of the following inclusion criteria:

* Normal, healthy male and female children and adults.
* Age 12 to 40 years.
* Written and verbal informed consent must be obtained. Subjects age 12 to 17 (inclusive) must sign an assent for the study and a parent or a legal guardian must sign the informed consent (per FDA letter 8.21.07).
* Women of child-bearing potential must be non-pregnant and non-nursing, and must be willing to avoid pregnancy during the course of the study and during the menstrual cycle following completion of their participation in the study, adequate contraception is defined as regular use of any two of the following: oral, injectable contraceptives, condoms, spermicides, diaphragm, IUD, implantable and contraceptive patches. (oral contraceptives if used for at least three months and injectable contraceptives if used for at least 6 months)- prior to enrollment in the study, or abstinence.
* Have at least 20 inflammatory (papules and pustules) and 25 non-inflammatory (open and closed comedones) lesions with a maximum of 2 nodulocystic lesions on the face (per FDA letter 8.21.07).
* Global severity score from 2-4
* Able to refrain from the use of all other topical acne medications or antibiotics during the treatment period.
* Considered reliable and capable of understanding their responsibility and role in the study.

Exclusion Criteria

A subject will be eligible to participate if they meet none of the following exclusion criteria:

* Subjects with active cystic acne as evidenced by more than 2 facial nodules.
* More than 40 papules and/or pustules (inflammatory lesions)
* More than 60 open and or closed comedones/milia (non-inflammatory lesions)
* Overall severity grade of less than 2 or greater than 4,
* History of allergy or hypersensitivity to tretinoin.
* Significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, or renal disease
* Use of systemic retinoid treatment within six months prior to study initiation.
* Oral contraceptives should not be started or changed within 3 months prior to study initiation or planned to change during the study.
* Pregnant or breast-feeding.
* Participation in a clinical study for acne within 4 months preceding study initiation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 958 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Cunningham, MD, Study Director — Cu-Tech
Locations (1):
- Cu-Tech, LLC, Mountain Lakes, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Generic: active cream
  Tretinoin: Topical skin
- Placebo: placebo cream
  Tretinoin: Topical skin
  placebo
- Brand: Tretinoin: Topical skin
Period: Overall Study
Arm/Group | Active Generic | Placebo | Brand
Started | 401 | 135 | 404
Completed | 318 | 110 | 337
Not Completed | 83 | 25 | 67

BASELINE CHARACTERISTICS:
Groups:
- Active Generic: Active generic group
- Brand: Brand group
- Placebo: Placebo group
- Total: Total of all reporting groups
Arm/Group | Active Generic | Brand | Placebo | Total
Number analyzed (Participants) | 401 | 404 | 135 | 940
Age, Continuous [Median (Standard Deviation); unit: years] | 17.2 (6.2) | 17.1 (6.1) | 17.6 (6.3) | 17.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 211 | 80 | 484
  Male | 208 | 193 | 55 | 456
Region of Enrollment [Number; unit: participants]
  United States | 401 | 404 | 135 | 940

OUTCOME MEASURES:

1. Primary Outcome: Acne Lesion Percent Reduction
Description: Reduction in number of Acne lesions by counting over 12 weeks
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: percent reduction of number of lesions
Arm/Group | Active Generic | Placebo | Brand
Number analyzed (Participants) | 318 | 110 | 337
percent reduction of number of lesions | -54.3 (10) | -35 (8) | -53.5 (10)

ADVERSE EVENTS:
Arm/Group | Active Generic | Placebo | Brand
Serious Adverse Events (participants affected / at risk) | 1/401 | 0/135 | 1/404
Other Adverse Events (participants affected / at risk) | 0/401 | 0/135 | 0/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Generic (N=401) | Placebo (N=135) | Brand (N=404)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — appendicitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other